CLINICAL TRIAL: NCT02105428
Title: Potential Impact of Polycystic Ovarian Syndrome on Protein Modifications and Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-007006
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Insulin Resistance; Overweight; Obese
Keywords: Polycystic Ovarian Syndrome (PCOS); Insulin Resistance; Overweight, Obese Women; Protein Metabolism; Post Translational Modifications
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary Control (No Intervention): Participants will be randomized to an exercise training program or sedentary control group. The sedentary will not perform any structured physical activity or exercise. Participants will be encouraged to maintain their sedentary lifestyle and will be monitored by an accelerometer to track physical activity.
- Aerobic Exercise Training (Experimental): Participants will perform 12-weeks of aerobic exercise training
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — A progressive increase in duration, frequency and intensity so the last 8 weeks of exercise are performed for 60 min, 5 days per week and at 80% of aerobic capacity. The duration includes a 5 minute warm up and 5 minute cool down. All exercise will be performed on a stationary bicycle (i.e., cycle ergometer).
  Arms: Aerobic Exercise Training

SUMMARY:
A goal of this study is to use a novel methodology to determine whether insulin resistance in women with polycystic ovary syndrome (PCOS) is related to the accumulation of proteins with modifications. This could lead to future research to determine if these modifications interfere with their proper function. Additionally, the investigators will determine how protein quality is affected by exercise training. Aerobic exercise enhances the endogenous oxidant buffering systems which may minimize oxidative damage to proteins. The investigators propose that aerobic exercise minimizes the accrual of modified proteins by increasing the synthesis of new proteins, but also by increasing the degradation and removal of old and damaged proteins. Based on our previous studies the investigators observed that insulin affects plasma protein synthesis and aerobic exercise improves insulin sensitivity not only in muscle but also in liver. The investigators therefore propose that aerobic exercise and related increase in insulin sensitivity (and decline in insulin levels) will reduce accumulation of old and modified skeletal muscle and plasma proteins leading to improved function.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 25 kg/m2 and 40 kg/m2
2. Fasting blood glucose < 126 mg/dL
3. Diagnosed with PCOS as outlined by the Rotterdam criteria
4. Insulin resistant as determined by a 3 hour oral glucose tolerance test

Exclusion Criteria:

1. Serum creatinine ≥1.5 mg/ dL.
2. Serum transaminase elevation ≥ 3 times the upper limit of normal range
3. Use of systemic glucocorticoids
4. Use of oral anticoagulation
5. Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Measured before and after 12 weeks
  To determine the effect of 12 weeks of aerobic exercise training or sedentary behavior on insulin sensitivity measured by a 3 hour hyperinsulinemic-euglycemic clamp and response to a mixed-meal.

SECONDARY OUTCOMES:
Protein modifications and accumulation | Before and after 12 weeks
  Alterations in protein modifications and accumulation will be measured by a novel methodology developed within our laboratory. Infusion of stable amino acid isotopes will be used to measure the accumulation of proteins before and after 12 weeks of aerobic exercise training or sedentary behavior. Plasma and muscle will be resolved using a two dimensional gel electrophoresis which will allow the identification of protein modifications and age.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States